CLINICAL TRIAL: NCT06329505
Title: National Taipei University of Nursing and Health Science
Brief Title: Impact of Extracorporeal Membrane Oxygenation Care Strategy Application Development
Status: Active, not recruiting | Type: Observational
Sponsor: Pei-Hung Liao (Other)
Responsible Party: Sponsor-Investigator, Pei-Hung Liao, Associate Professor, National Taipei University of Nursing and Health Sciences
Organization: National Taipei University of Nursing and Health Sciences (Other)
Other Study IDs: 111-085-B
Record Dates: First submitted 2024-03-13; First posted 2024-03-26 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Learning Problem
Keywords: Learning

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of this study was to develop an educational training App for ECMO care, and to apply a blended learning approach to improve the knowledge and skills of nurses.

DETAILED DESCRIPTION:
In recent years, for patients with acute cardiac infarction, severe cardiac shock, and refractory acute respiratory distress syndrome, the intervention of Extracorporeal Membrane Oxygenation (ECMO) has become an adjunctive treatment for severe cardiopulmonary diseases, which can temporarily replace cardiopulmonary function, slow the deterioration of cardiopulmonary function, and buy time to assist in clinical treatment. However, the education and training of ECMO is mainly based on traditional classroom teaching, which has also been affected by COVID-2019, resulting in training process difficulties as nurses are easily restricted by time and environment.

ELIGIBILITY:
Inclusion Criteria:

* licensed nurse practitioners working in the intensive care center of the teaching hospital and willing to participate in the study.

Exclusion Criteria:

* those who did not use smart phones.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: There was a total of 97 participants in this study, with an average of 9 years of nursing experience; the shortest experience was 1 year, and the longest was 29 years, of which 35 (36%) participants were nurses with less than 5 years of experience, and 36 (37%) were nurses with more than 10 years of experience.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Comparison of knowledge and skills of nurses between groups after the intervention For 6 months. | 6 months
  The instruments of this study included a questionnaire survey, the development of the ECMO Care Strategy App, and a blended learning design. The questionnaire survey consisted of three parts: the first part was the basic attributes, the second part was the perception of the ECMO knowledge and care behaviors, and the third part was the ECMO Care Strategy App System Usability Assessment Scale. The questionnaire content was based on the ECMO training literature and digital learning of Rouleau et al. (2019), Thomas et al. (2019), Chaves et al. (2019), Jiritano et al. (2020), as well as the content of the in-hospital ECMO education and training manual, including the care knowledge and perception of care behaviors, for a total of 18 questions.

CONTACTS AND LOCATIONS:
Overall Officials: Pei-Hung Liao, PH.D., Study Director — National Taipei university of nursing and health science
Locations (1):
- National Taipei university of nursing and health science, Taipei, Taiwan